CLINICAL TRIAL: NCT05690529
Title: Echocardiographic Markers of Atrial Fibrillation Recurrence Post Radiofrequency Ablation
Acronym: Echo-If-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, Diogo de Almeida Fernandes, Dr., Unidade Local de Saúde de Coimbra, EPE
Other Study IDs: Echo AF 2021
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No recurrence: No recurrence of AF
  Interventions: Procedure: Ablation
- Recurrence: Recurrence of AF
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation — Radiofrequency AF ablatoon

SUMMARY:
Determine echocardiographic predictors of atrial fibrillation recurrence post radiofrequency Ablation and evaluate markers of low voltage areas on 3D mapping.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal or persistent ablation

Exclusion Criteria:

* previous AF ablation
* previous left atrial ablation
* refusal to give informed consent
* congenital cradiomiopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radiofrequency AF ablation guided by 3D mapping
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 1 year

SECONDARY OUTCOMES:
Low voltage areas | At procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided